CLINICAL TRIAL: NCT00033709
Title: A Phase II Study of Combination Therapy of a Protracted Oral Schedule of Temozolomide and Thalidomide as First-Line or Subsequent Therapy for Patients With Metastatic, Locally Advanced or Unresectable Leiomyosarcoma
Brief Title: Temozolomide and Thalidomide in Treating Patients With Metastatic, Locally Advanced, or Unresectable Leiomyosarcoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Herbert Irving Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000069314; CPMC-IRB-14323; NCI-G02-2060
Record Dates: First submitted 2002-04-09; First posted 2003-01-27 (Estimated); Last update posted 2014-01-06 (Estimated); Status verified 2005-05

CONDITIONS: Sarcoma
Keywords: adult leiomyosarcoma; stage III adult soft tissue sarcoma; recurrent adult soft tissue sarcoma; stage III uterine sarcoma; stage IV uterine sarcoma; recurrent uterine sarcoma; uterine leiomyosarcoma; stage IV adult soft tissue sarcoma
MeSH Terms: conditions — Sarcoma; Leiomyosarcoma | interventions — Temozolomide; Thalidomide

INTERVENTIONS:
Drug: temozolomide
Drug: thalidomide

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Thalidomide may stop the growth of cancer by stopping blood flow to the tumor. Combining temozolomide with thalidomide may kill more tumor cells.

PURPOSE: Phase II trial to study the effectiveness of combining temozolomide with thalidomide in treating patients who have metastatic, locally advanced, or unresectable leiomyosarcoma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the efficacy of temozolomide and thalidomide in patients with metastatic, locally advanced, or unresectable leiomyosarcoma.
* Determine the time to progression in patients treated with this regimen.
* Determine the overall survival of patients treated with this regimen.
* Determine the clinical and laboratory toxic effects and tolerability of this regimen in these patients.

OUTLINE: Patients receive oral temozolomide once daily for 7 days every other week and oral thalidomide once daily. Treatment continues for up to 26 weeks in the absence of disease progression or unacceptable toxicity.

PROJECTED ACCRUAL: A total of 15-25 patients will be accrued for this study within 7.5-25 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed leiomyosarcoma

  * Metastatic, locally advanced, or unresectable
* Ineligible for other high priority national or institutional study
* At least 1 unidimensionally measurable lesion documented on radiologic study

  * At least 2 cm by 2 cm
  * Not previously irradiated unless disease progression at the site is evident
* No brain metastases

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* SWOG 0-2

Life expectancy:

* More than 2 months

Hematopoietic:

* WBC greater than 3,000/mm^3
* Neutrophil count at least 1,500/mm^3
* Platelet count greater than 70,000/mm^3
* Hemoglobin at least 10 g/dL

Hepatic:

* Bilirubin less than upper limit of normal (ULN)
* SGOT or SGPT less than 1.5 times ULN*
* Alkaline phosphatase less than 2 times ULN* NOTE: * Less than 5 times ULN if documented liver disease

Renal:

* Creatinine less than 1.5 times normal OR
* Creatinine clearance greater than 60 mL/min
* BUN less than 1.5 times normal

Other:

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use 2 forms of effective contraception for 4 weeks before, during, and for 4 weeks after study therapy
* No acute infection requiring systemic antibiotics
* No frequent vomiting or medical condition that would preclude intake of oral medication (e.g., partial bowel obstruction)
* No other serious medical or psychiatric illness that would preclude study participation
* No prior malignancy except curatively treated carcinoma in situ of the cervix or skin cancer

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* At least 4 weeks since prior chemotherapy
* No more than 3 prior systemic chemotherapy regimens for metastatic, locally advanced, or unresectable leiomyosarcoma
* Prior dacarbazine allowed

Endocrine therapy:

* Not specified

Radiotherapy:

* See Disease Characteristics
* At least 4 weeks since prior radiotherapy
* No prior radiotherapy to 50% or more of bone marrow
* Concurrent radiotherapy for local control or palliative therapy for painful bony or soft tissue lesion allowed

Surgery:

* At least 4 weeks since prior surgery and recovered

Other:

* Recovered from all prior therapies
* No other concurrent investigational drugs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2002-03

PRIMARY OUTCOMES:
Response (complete and partial response)

SECONDARY OUTCOMES:
Time to progression
Overall survival
Clinical benefit

CONTACTS AND LOCATIONS:
Overall Officials: Robert N. Taub, MD, PhD, Study Chair — Herbert Irving Comprehensive Cancer Center
Locations (1):
- Herbert Irving Comprehensive Cancer Center at Columbia University, New York, New York, United States

REFERENCES:
- [Result] Boyar MS, Hesdorffer M, Keohan ML, Jin Z, Taub RN. Phase II Study of Temozolomide and Thalidomide in Patients with Unresectable or Metastatic Leiomyosarcoma. Sarcoma. 2008;2008:412503. doi: 10.1155/2008/412503. Epub 2008 Nov 16. PMID 19043564